CLINICAL TRIAL: NCT03474679
Title: A Phase 3 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib in Subjects With Steroid Dependent/Refractory Chronic Graft Versus Host Disease (cGVHD)
Brief Title: A Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib in Participants With Steroid Dependent/Refractory Chronic Graft Versus Host Disease (cGVHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108443; 54179060GVH3001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ibrutinib (Experimental): Participants will receive 420 milligram (mg) oral ibrutinib once daily starting on Week 1 Day 1, unless they have intervening unacceptable toxicity or meet other criteria for participants discontinuation.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Participants will receive 420 mg (3 * 140 mg capsules) oral ibrutinib once daily starting on Week 1 Day 1, unless they have intervening unacceptable toxicity or meet other criteria for participants discontinuation.
  Other Names: PCI-32765; JNJ-54179060

SUMMARY:
The purpose of this study is to evaluate efficacy of ibrutinib in Japanese participants with steroid dependent/refractory chronic graft versus host disease (cGVHD) by measuring overall cGVHD response (complete response [CR] and partial response [PR] defined by National Institutes of Health [NIH] consensus development project criteria [2014]).

ELIGIBILITY:
Inclusion Criteria:

* Steroid dependent/refractory chronic graft versus host disease (cGVHD) defined as modified National Institutes of Health (NIH) criteria (2014) below at any time post-hematopoietic cell transplant (post-HCT): a) Dependent disease, defined as, when glucocorticoid (prednisolone doses greater than or equal to [>=] 0.25 milligram per kilogram per day (mg/kg/day)or >=0.5 milligram per kilogram (mg/kg) every other day) are needed to prevent recurrence or progression of manifestations as demonstrated by unsuccessful attempts to taper the dose to lower levels on at least 2 occasions, separated by at least 8 weeks. In case of inability to taper the dose to less than or equal to (<=)0.25 mg/kg/day or <=0.5 mg/kg every other day (prednisolone doses) due to recurrence or progression of cGVHD manifestations, it is considered as steroid-dependent disease if the lowest tapering dose of the second occasion is equal or higher than the lowest tapering dose of the first occasion; b) Refractory disease, defined as, when cGVHD manifestations progress despite the use of a regimen containing glucocorticoid (prednisolone at >=1 mg/kg/day for at least 1 week) or persist without improvement despite continued treatment with glucocorticoid (prednisolone at >=0.5 mg/kg/day or 1 mg/kg every other day) for at least 4 weeks
* Participants must be receiving baseline systemic glucocorticoid therapy for cGVHD at study entry. The dose of steroids must be stable for 14 days prior to starting ibrutinib
* At the time of trial enrollment, participants may be receiving other immunosuppressive therapies in addition to glucocorticoids. Immunosuppressant doses must be stable for 14 days prior to starting ibrutinib
* Clinically stable or worsening cGVHD for a minimum of 14 days between screening and Day 1 cGVHD response assessment
* Karnofsky or Lansky (participants less than [<]16 years) performance status >=60

Exclusion Criteria:

* Active acute graft versus host disease (GVHD)
* More than 3 previous systemic treatments for cGVHD. Treatment with glucocorticoids is considered a treatment for cGVHD and should be included in determining the number of previous treatments
* History of treatment with a tyrosine kinase inhibitor (example [e.g.] imatinib), purine analogs, or other cancer chemotherapy in the 4 weeks prior to starting ibrutinib. Participants may have received ibrutinib pre-transplant for other reasons besides cGVHD such as for the treatment of leukemia or lymphoma
* History of treatment with monoclonal T and B cell antibodies in the 8 weeks prior to starting ibrutinib
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of ibrutinib

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (15):
- Japan (15):
  - Anjo Kosei Hospital, Anjo-shi
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō City
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Tokai University Hospital, Isehara
  - Osaka Women's and Children's Hospital, Izumi
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Okayama University Hospital, Okayama
  - Osaka City University Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - National Center for Child Health and Development, Setagaya Ku

REFERENCES:
- [Derived] Toyosaki M, Doki N, Shiratori S, Osumi T, Okada M, Kawakita T, Sawa M, Ishikawa T, Ueda Y, Hatayama T, Yoshinari N, Fujikawa E. Long-term Use of Ibrutinib in Japanese Patients with Steroid Dependent/Refractory cGVHD: Final Analysis of Multicenter Study. Blood Cell Ther. 2023 Nov 10;6(4):104-113. doi: 10.31547/bct-2023-010. eCollection 2023 Nov 25. PMID 38149026
- [Derived] Doki N, Toyosaki M, Shiratori S, Osumi T, Okada M, Kawakita T, Sawa M, Ishikawa T, Ueda Y, Yoshinari N, Nakahara S. An Open-Label, Single-Arm, Multicenter Study of Ibrutinib in Japanese Patients With Steroid-dependent/Refractory Chronic Graft-Versus-Host Disease. Transplant Cell Ther. 2021 Oct;27(10):867.e1-867.e9. doi: 10.1016/j.jtct.2021.05.019. Epub 2021 Jun 6. PMID 34102349

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib 420 mg: Participants with steroid dependent/refractory chronic graft versus host disease (cGVHD) received ibrutinib 420 milligrams (mg) (3*140 mg capsule) orally once daily on Week 1 Day 1 until participants had intervening unacceptable toxicity or met other criteria for discontinuation.
Period: Overall Study
Arm/Group | Ibrutinib 420 mg
Started | 19
Completed | 11
Not Completed | 8
Not completed — Death | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (16.24)
Age, Customized [Count of Participants; unit: Participants]
  Less Than or Equal to 17 years (adolescent) | 1
  From 18 to 64 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve complete response (CR) or partial response (PR) in the absence of new therapy for chronic graft versus host disease (cGVHD) and absence of progression of underlying disease or death based on the National Institutes of Health (NIH) Consensus Development Project Criteria (2014). CR is defined as resolution of all manifestations in each organ or site; PR is defined as improvement in at least 1 organ or site without progression in any other organ or site; and chronic graft versus host disease (cGVHD) progression is defined as clinically meaningful worsening in 1 or more organs regardless of improvement in other organs.
Time Frame: Up to 3 year 6 months
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Percentage of participants | 84.2

2. Secondary Outcome: Sustained Response Rate
Description: Sustained response rate was defined as percentage of participants with NIH defined CR or PR that was sustained for at least 20 weeks. CR is defined as resolution of all manifestations in each organ or site; PR is defined as improvement in at least 1 organ or site without progression in any other organ or site.
Time Frame: Up to 3 year 6 months
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug and achieved PR or better response.
Measure: Number; unit: Percentage of participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 16
Percentage of participants | 68.8

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the duration from the date of initial response (CR or PR) to the date of progressive cGVHD or death, whichever occurred first. CR is defined as resolution of all manifestations in each organ or site; PR is defined as improvement in at least 1 organ or site without progression in any other organ or site; and cGVHD progression is defined as clinically meaningful worsening in 1 or more organs regardless of improvement in other organs.
Time Frame: Up to 3 year 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 16
Months | NA [5.30 to NA] — Here, 'NA' indicates that median and upper limit of 95% confidence interval were not estimable due to the less number of events.

4. Secondary Outcome: cGVHD Response Rate at Each Timepoints
Description: cGVHD response rate was defined as percentage of participants with NIH defined CR or PR at each timepoint. CR is defined as resolution of all manifestations in each organ or site; PR is defined as improvement in at least 1 organ or site without progression in any other organ or site.
Time Frame: Weeks 5, 13, 25, 37, 49, 61, 73, 85, 97, 109, 121, 133, 145, 157
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Percentage of participants
  Week 5 | 26.3 [9.1 to 51.2]
  Week 13 | 42.1 [20.3 to 66.5]
  Week 25 | 52.6 [28.9 to 75.6]
  Week 37 | 47.4 [24.4 to 71.1]
  Week 49 | 47.4 [24.4 to 71.1]
  Week 61 | 42.1 [20.3 to 66.5]
  Week 73 | 36.8 [16.3 to 61.6]
  Week 85 | 31.6 [12.6 to 56.6]
  Week 97 | 31.6 [12.6 to 56.6]
  Week 109 | 31.6 [12.6 to 56.6]
  Week 121 | 36.8 [16.3 to 61.6]
  Week 133 | 31.6 [12.6 to 56.6]
  Week 145 | 26.3 [9.1 to 51.2]
  Week 157 | 10.5 [1.3 to 33.1]

5. Secondary Outcome: Change in the Amount of Corticosteroid Required Over Time
Description: Change in the amount of corticosteroid required over time was reported.
Time Frame: Baseline, Weeks 24, 48, 96, and 144
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug. Here, 'n' (number analyzed) represents number of participants evaluable at the specified timepoints.
Measure: Median (Full Range); unit: Milligrams per kilograms per day
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Milligrams per kilograms per day
  Baseline | 0.270 [0.08 to 1.77]
  Week 24: number analyzed (Participants) | 13
  Week 24 | 0.250 [0.08 to 0.87]
  Week 48: number analyzed (Participants) | 11
  Week 48 | 0.150 [0.06 to 0.64]
  Week 96: number analyzed (Participants) | 9
  Week 96 | 0.140 [0.01 to 0.59]
  Week 144: number analyzed (Participants) | 4
  Week 144 | 0.140 [0.05 to 0.56]

6. Secondary Outcome: Percentage of Participants With Overall Improvement in Lee cGVHD Symptom Scale Score
Description: Percentage of participants with overall improvement in Lee cGVHD symptom scale score was reported. Lee cGVHD symptom scale is a patient-reported symptom scale used to measure symptom burden and has 7 subscales (Skin, Eyes and Mouth, Breathing, Eating and Digestion, Muscles and Joints, Energy, and Mental and Emotional) with ratings as follows: 0-Not at all, 1-Slightly, 2-Moderately, 3-Quite a bit, 4-Extremely, with lower values representing a better outcome. A score was calculated for each subscale by taking the mean of all items completed if more than 50% were answered and normalizing to a 0 to 100 with a higher score indicating worse symptoms. An overall score was calculated as the average of these 7 subscales if at least 4 subscales had valid scores. A change of greater than or equal to (>=) 7 points on the Lee cGVHD symptom scale overall score was considered significant and relates to improvement in quality of life (QoL).
Time Frame: Up to 3 year 6 months
Population: All treated analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Percentage of participants | 52.6 [28.9 to 75.6]

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs are adverse events with onset during the treatment phase or that were a consequence of a preexisting condition that has worsened since baseline, and occurred during treatment or within 30 days following the last dose of study treatment, or any adverse event that was considered study treatment-related regardless of the start date of the event.
Time Frame: Up to 3 year 6 months
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Participants | 19

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Measurable Concentration (AUC [0-last]) of Ibrutinib
Description: AUC(0-last) is defined as area under the plasma concentration-time curve from time zero to time of last measurable concentration of ibrutinib.
Time Frame: Day 1 of Weeks 1 and 2
Population: The pharmacokinetic (PK) evaluable analysis set included all enrolled participants who received at least one dose of study drug and had at least 1 postdose PK sample obtained.
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
hours*nanograms per milliliter (h*ng/mL)
  Week 1: Day 1 | 3683.7 (3146.9)
  Week 2: Day 1 | 4024.8 (4287.2)

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC [0-24]) of Ibrutinib
Description: AUC(0-24) is defined as area under the plasma concentration-time curve from time zero to 24 hours of ibrutinib.
Time Frame: 0 to 24 hours (Day 1 of Weeks 1 and 2)
Population: The PK evaluable analysis set included all enrolled participants who received at least one dose of study drug and had at least 1 postdose PK sample obtained. Here, 'n' (number analyzed) represents number of participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
hour*ng/mL
  Week 1: Day 1: number analyzed (Participants) | 7
  Week 1: Day 1 | 2929.3 (1797.4)
  Week 2: Day 1 | 4035.6 (4277.2)

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ibrutinib
Description: Cmax is defined as maximum observed plasma concentration of ibrutinib.
Time Frame: Day 1 of Weeks 1 and 2
Population: The PK evaluable analysis set included all enrolled participants who received at least one dose of study drug and had at least 1 postdose PK sample obtained.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Nanograms per milliliter (ng/mL)
  Week 1: Day 1 | 490.45 (366.07)
  Week 2: Day 1 | 478.01 (508.08)

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Ibrutinib
Description: Tmax is defined as time to reach the maximum observed plasma concentration of ibrutinib.
Time Frame: Day 1 of Weeks 1 and 2
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Hours
  Week 1: Day 1 | 3.87 [1.78 to 5.75]
  Week 2: Day 1 | 4.02 [1.75 to 5.43]

12. Secondary Outcome: Elimination Half-Life (t1/2) of Ibrutinib
Description: T1/2 is defined as elimination half-life of ibrutinib.
Time Frame: Day 1 of Weeks 1 and 2
Population: The PK evaluable analysis set included all enrolled participants who received at least one dose of study drug and had at least 1 postdose PK sample obtained. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Hours
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 4
Hours
  Week 1: Day 1 | 4.9 [4.4 to 5.2]
  Week 2: Day 1 | 4.4 [3.8 to 10.2]

13. Secondary Outcome: Apparent Clearance (CL/F) of Ibrutinib
Description: CL/F is defined as apparent clearance of ibrutinib.
Time Frame: Day 1 of Weeks 1 and 2
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliters per hour (mL/h)
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 4
Milliliters per hour (mL/h)
  Week 1: Day 1 | 194211 (106164)
  Week 2: Day 1 | 162457 (31966)

14. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Ibrutinib
Description: Vd/F is defined as apparent volume of distribution of ibrutinib.
Time Frame: Day 1 of Weeks 1 and 2
Population: The PK evaluable analysis set included enrolled participants who received at least one dose of study drug and had at least 1 postdose PK sample obtained. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 4
Milliliters (mL)
  Week 1: Day 1 | 1350160 (748511)
  Week 2: Day 1: number analyzed (Participants) | 0

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Ibrutinib
Description: AUC(0-infinity) is defined as area under the plasma concentration-time curve from time zero to infinite time of ibrutinib.
Time Frame: Day 1 of Weeks 1 and 2
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 4
hour*ng/mL
  Week 1: Day 1 | 2643.8 (1656.2)
  Week 2: Day 1 | 2659.2 (506.57)

16. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Measurable Concentration (AUC [0-last]) of PCI-45227
Description: AUC(0-last) is defined as area under the plasma concentration-time curve from time zero to time of last measurable concentration of PCI-45227.
Time Frame: Day 1 of Weeks 1 and 2
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
h*ng/mL
  Week 1: Day 1 | 1976.9 (968.83)
  Week 2: Day 1 | 2547.6 (999.00)

17. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC [0-24]) of PCI-45227
Description: AUC(0-24) is defined as area under the plasma concentration-time curve from time zero to 24 hours of PCI-45227.
Time Frame: 0 to 24 hours (Day 1 of Weeks 1 and 2)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
hour*ng/mL
  Week 1: Day 1: number analyzed (Participants) | 6
  Week 1: Day 1 | 1803.0 (585.84)
  Week 2: Day 1 | 2547.6 (999.00)

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PCI-45227
Description: Cmax is defined as maximum observed plasma concentration of PCI-45227.
Time Frame: Day 1 of Weeks 1 and 2
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
ng/mL
  Week 1: Day 1 | 185.37 (91.874)
  Week 2: Day 1 | 203.16 (82.292)

19. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PCI-45227
Description: Tmax is defined as time to reach the maximum observed plasma concentration of PCI-45227.
Time Frame: Day 1 of Weeks 1 and 2
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 19
Hours
  Week 1: Day 1 | 4.00 [1.88 to 6.18]
  Week 2: Day 1 | 4.02 [0.00 to 5.28]

20. Secondary Outcome: Elimination Half-Life (t1/2) of PCI-45227
Description: T1/2 is defined as elimination half-life of PCI-45227.
Time Frame: Day 1 of Weeks 1 and 2
Population: The PK evaluable analysis set is defined as all enrolled participants who received at least one dose of study drug and had at least 1 postdose PK sample obtained. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants who were evaluable for specified timepoints.
Measure: Median (Full Range); unit: Hours
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 4
Hours
  Week 1: Day 1 | 5.9 [5.2 to 6.5]
  Week 2: Day 1: number analyzed (Participants) | 1
  Week 2: Day 1 | 5.4 [5.4 to 5.4]

21. Secondary Outcome: Apparent Clearance (CL/F) of PCI-45227
Description: CL/F is defined as apparent clearance of PCI-45227.
Time Frame: Day 1 of Weeks 1 and 2
Population: The PK evaluable analysis set included all enrolled participants who received at least one dose of study drug and had at least 1 postdose PK sample obtained. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure and 'n' (number analyzed) represents number of participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 4
mL/h
  Week 1: Day 1 | 251681 (68392)
  Week 2: Day 1: number analyzed (Participants) | 1
  Week 2: Day 1 | 111922 (NA) — Here, 'NA' indicates that standard deviation could not be calculated for a single participant.

22. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of PCI-45227
Description: Vd/F is defined as apparent volume of distribution of PCI-45227.
Time Frame: Day 1 of Weeks 1 and 2
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 4
mL
  Week 1: Day 1 | 2148283 (653626)
  Week 2: Day 1: number analyzed (Participants) | 0

23. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of PCI-45227
Description: AUC(0-infinity) is defined as area under the plasma concentration-time curve from time zero to infinite time of PCI-45227.
Time Frame: Day 1 of Weeks 1 and 2
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Ibrutinib 420 mg
Number analyzed (Participants) | 4
hour*ng/mL
  Week 1: Day 1 | 1766.1 (478.74)
  Week 2: Day 1: number analyzed (Participants) | 1
  Week 2: Day 1 | 3752.6 (NA) — Here, 'NA' indicates that standard deviation could not be calculated for a single participant.

ADVERSE EVENTS:
Time Frame: Up to 3 year 6 months
Description: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Ibrutinib 420 mg
All-Cause Mortality (participants affected / at risk) | 7/19
Serious Adverse Events (participants affected / at risk) | 12/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib 420 mg (N=19)
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 1
Liver Disorder (Hepatobiliary disorders) | 1
Anaphylactic Reaction (Immune system disorders) | 1
Appendiceal Abscess (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Covid-19 (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pneumonia Bacterial (Infections and infestations) | 1
Pneumonia Fungal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Atypical Femur Fracture (Injury, poisoning and procedural complications) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1
Renal Impairment (Renal and urinary disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib 420 mg (N=19)
Anaemia (Blood and lymphatic system disorders) | 3
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 1
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 2
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Splenic Infarction (Blood and lymphatic system disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiac Failure Chronic (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Cataract (Eye disorders) | 4
Conjunctival Erosion (Eye disorders) | 1
Conjunctival Hyperaemia (Eye disorders) | 1
Dry Eye (Eye disorders) | 2
Glaucoma (Eye disorders) | 2
Ocular Hypertension (Eye disorders) | 1
Photophobia (Eye disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Dental Caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Enterocolitis (Gastrointestinal disorders) | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 1
Gastric Mucosal Hypertrophy (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 9
Tooth Loss (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Generalised Oedema (General disorders) | 2
Malaise (General disorders) | 2
Oedema Peripheral (General disorders) | 4
Physical Deconditioning (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Liver Disorder (Hepatobiliary disorders) | 1
Food Allergy (Immune system disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 1
Seasonal Allergy (Immune system disorders) | 1
Appendiceal Abscess (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 6
Conjunctivitis (Infections and infestations) | 3
Cytomegalovirus Infection (Infections and infestations) | 1
Haematoma Infection (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Oral Candidiasis (Infections and infestations) | 1
Otitis Externa (Infections and infestations) | 1
Paronychia (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia Aspiration (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Pneumonia Fungal (Infections and infestations) | 1
Postoperative Wound Infection (Infections and infestations) | 1
Pseudomembranous Colitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 6
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1
Atypical Femur Fracture (Injury, poisoning and procedural complications) | 1
Bone Contusion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Joint Injury (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 2
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Amylase Increased (Investigations) | 1
Aspergillus Test Positive (Investigations) | 1
Blood Beta-D-Glucan Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 2
Blood Fibrinogen Decreased (Investigations) | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1
Haemoglobin Decreased (Investigations) | 1
Lipase Increased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 2
Platelet Count Decreased (Investigations) | 6
Weight Decreased (Investigations) | 2
Weight Increased (Investigations) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Lipid Metabolism Disorder (Metabolism and nutrition disorders) | 1
Zinc Deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Immobilisation Syndrome (Musculoskeletal and connective tissue disorders) | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Acute Lymphocytic Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 1
Intercostal Neuralgia (Nervous system disorders) | 1
Restless Legs Syndrome (Nervous system disorders) | 1
Toxic Encephalopathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 2
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2
Drug Eruption (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 2
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Purpura (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin Induration (Skin and subcutaneous tissue disorders) | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT03474679/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT03474679/SAP_001.pdf